CLINICAL TRIAL: NCT02511899
Title: Investigation of the Influence of Careless™, a Mangifera Indica Fruit Powder, on Microcirculation and Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital Solutions Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BTS850/15
Record Dates: First submitted 2015-07-22; First posted 2015-07-30 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Microcirculation; Metabolism; Cardiovascular Disease
Keywords: Microcirculation; Endothelial function; Metabolism; Cardiovascular Disease; human study; healthy subjects; Mangifera indica; Careless
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mango fruit powder 100mg (Active Comparator): Mango fruit powder 100mg
  Interventions: Dietary Supplement: Mango fruit powder
- Mango fruit powder 300mg (Active Comparator): Mango fruit powder 300mg
  Interventions: Dietary Supplement: Mango fruit powder

INTERVENTIONS:
Dietary Supplement: Mango fruit powder — Dietary supplement; Mango fruit powder
  Other Names: Careless

SUMMARY:
Investigation of the acute effects of a single dose of Careless™, a Mangifera indica fruit powder on cutaneous microcirculation and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Subject is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry and haematology
* Healthy normal skin condition at the forearm
* BMI: 19-30 kg/m2
* Female
* Age ≥ 40 and ≤ 70 years
* Nonsmoker
* Able and willing to follow the study protocol procedures

Exclusion Criteria:

* Relevant history, presence of any medical disorder or chronic intake of medication/dietary supplements (e.g. polyphenols, L-Arginine, Niacin, medication of haemodilution, blood flow stimulating products like Aspirin) potentially interfering with this study at screening
* For this study clinically relevant abnormal laboratory, vital signs or physical findings at screening
* Atopic dermatitis or affected skin at the forearm
* Regular consumption of caffeine > 275 mg (equivalent to 3-4 cups of coffee or 9 cups of black tea)
* Change of dietary habits within the 2 weeks prior to screening (for instance start of a diet high in vegetables and fruits (≥ 5 portions per day))
* Diet high in vegetables and fruits ≥ 5 portions per day
* Participants anticipating a change in their lifestyle or physical activity levels since this may also influence the results
* Subjects not willing to avoid polyphenol rich foods and abstain from beverages containing caffeine the day prior to visit 1 and 2
* Subjects not willing to abstain from intake of analgesic medication (e.g. Aspirin) 24 hours prior to and during visit 1 and 2
* Sunbathing or the use of sun-beds 2 weeks prior to study days
* Injury on the finger, influencing the EndoPAT™ measurement
* Subjects with history of drug, alcohol or other substances abuse, or other factors limiting their ability to co-operate during the study
* Known hypersensitivity to the study product or to single ingredients
* Pregnant subject or subject planning to become pregnant during the study; breast-feeding subject.
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 4 weeks prior to visit 1 or during the study
* Subject involved in any clinical or food study within the preceding month

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Delta change of dermal microcirculation before and after intake (1h, 2h, 3h, 4h and 6h post) measured by O2C technology | baseline before intake at the same day and 1hour, 2hour, 3hour, 4hour and 6hour post intake
  Change over time for microcirculation
Delta change of endothelial function using EndoPAT™ (baseline and 3hour post) | baseline before intake at the same day and 3 hours post intake
  Changes over time of endothelial function

SECONDARY OUTCOMES:
Tolerability, number of participants with adverse events | after 6 hours of intake

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Reule, PhD, Study Director — BioTeSys GmbH
Locations (1):
- BioTeSys GmbH, Esslingen am Neckar, Germany